CLINICAL TRIAL: NCT00331747
Title: Three Dimensional Gait Evaluation in Relapsing Remitting Multiple Sclerosis Patients Treated With Glatiramer Acetate
Brief Title: Gait Evaluation in Multiple Sclerosis Patients Treated With Glatiramer Acetate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3985-UG-CTIL
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2006-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glatiramer Acetate

INTERVENTIONS:
Drug: Glatiramer acetate

SUMMARY:
Hypothesis: Treatment with Glatiramer acetate prevents deterioration of gait in multiple sclerosis (MS) patients.

During the study patients will undergo a 3 dimensional gait analysis before starting treatment with glatiramer acetate and after 1 year of treatment.

DETAILED DESCRIPTION:
Patients with a definite diagnosis of relapsing remitting multiple sclerosis (MS) will undergo a 3 dimensional gait analysis before initiation of treatment with glatiramer acetate. The gait analysis will include kinematic evaluation using a Charnwood Dynamics CODA CX-1 system, 4 AMTI force plates and a Noraxon telemetric EMG system. Patients will be videotaped and will also undergo a detailed physical examination by a physical therapist.

Treatment with Glatiramer acetate will be initiated after the gait analysis. Therapy will be observed and controlled by a neurologist fromn the staff of the Multiple Sclerosis Center.

Repeat gait analysis will be performed after one year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of multiple sclerosis
* EDSS less than 5.5
* No cognitive disability

Exclusion Criteria:

* EDSS over 5.5
* Inability to cooperate with gait analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-05

PRIMARY OUTCOMES:
Computerized gait analysis: at the beginning of treatment and after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Uri Givon, MD, Principal Investigator — Sheba Medical Center; Tel Aviv University; Anat Achiron, MD, PhD, Study Chair — Sheba Medical Center; Tel Aviv University
Locations (1):
- Multiple Sclerosis Center, Sheba Medical Center, Tel Litwinsky, Israel